CLINICAL TRIAL: NCT00797004
Title: Olfactory Dysfunction of Rhinosinusitis
Acronym: ODOR
Status: Completed | Type: Observational
Sponsor: Greg Davis (Other)
Responsible Party: Sponsor-Investigator, Greg Davis, Assistant Professor, University of Washington
Organization: University of Washington (Other)
Other Study IDs: 35031-B
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Rhinosinusitis
Keywords: olfactory dysfunction
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- endoscopic sinus procedure candidates

SUMMARY:
The purpose of this research is to improve understanding of the molecular and functional properties of the human olfactory system.

The specific aims are:

* to determine the location of AC3 and Golf proteins in the human olfactory epithelium from freshly harvested nasal/sinus tissue of surgical patients
* to perform objective functional studies on fresh human nasal/sinus tissue using an electro-olfactogram (EOG) whic measures the electrical activity of olfactory sensory neurons in fresh biopsied tissue in response to odor or pheromone stimulation. An organotypic culture system for human tissue has been established to optimize the electrical signal acquisition.
* to correlate the AC3 and Golf expression profiles with pre-operative testing of human olfactory function
* to correlate the EOG findings with pre-operative testing of human olfactory function.
* to systematically evaluate the role of individual intranasal agents on olfaction to further optimize the electrical signal acquisition from olfactory tissue.

DETAILED DESCRIPTION:
This is a prospective cohort study. Subjects will be recruited from the group of patients at the University of Washington Otolaryngology-Head and Neck Surgery Clinic who will undergo endoscopic sinus surgery for chronic sinusitis and other disorders of the nasal cavity and sinuses.

Subjects will sign consent and complete a subjective smell test (UPSIT--University of Pennsylvania Smell Identification Test), and the SNOT-20 (Sinonasal Outcome Test-20)

During their surgery, subjects will have two to four pieces of normally discarded tissue preserved for the study. Subjects will also have two to four pieces of healthy tissue removed (total size approximately that of a pencil eraser tip)depending on the type of surgery involved. The following procedures will be performed on these tissues:

* immunocytochemistry utilizing antibodies to AC3 and Golf to determine the patterns and levels of expression of these proteins
* two odorants, isoamyl acetate and citralva, to elicit odorant-induced activity from the human olfactory sensory neurons. The tissue will also be subjected to two putative human pheromones: 4,16-androstadiene-3-ol and 1,3,5(10),16-estrateraen-3-ol.
* application of six commonly used intranasal agents: 0.9% saline, 1:1000,000 epinephrine, 0.05% oxymetazoline, 1% lidocaine, Zicam (0.12% zinc gluconate) and Nasocort AQ (triamcinolone acetate).

ELIGIBILITY:
Inclusion Criteria:

* over 18 yrs. of age, scheduled for: a.) endoscopic sinus surgery for chronic sinusitis, b.) endoscopic transnasal approach to the pituitary for pituitary tumor removal, c.) endoscopic inferior turbinectomy for nasal congestion d.)endoscopic repair of cerebrospinal fluid leaks

Exclusion Criteria:

* unable to give informed consent or complete questionnaires due to language, cognitive impairment or sever medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical patients from the UW Otolaryngology - Head and Neck surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg E Davis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Lim JH, Davis GE, Rue TC, Storm DR. Human sinonasal explant system for testing cytotoxicity of intranasal agents. Int Forum Allergy Rhinol. 2012 Jan-Feb;2(1):63-8. doi: 10.1002/alr.20110. Epub 2011 Dec 13. PMID 22170775